CLINICAL TRIAL: NCT03517124
Title: Success and Survival of e.Max and KHF2 Etched Zirconia Cemented With Resin Cement - a Randomized Controlled Clinical Study
Brief Title: Ceramic Tooth Restorations - a Comparison Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oslo (Other)
Collaborators: Nordic Institute of Dental Materials (Unknown)
Responsible Party: Principal Investigator, Hans Jacob Rønold, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/957
Record Dates: First submitted 2017-12-29; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Zirconium oxide; surface treatment; resin cement

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia restorations (Experimental): Dental restorations in surface modified zirconia bonded to tooth substance by dual cure resin cement
  Interventions: Other: Ceramic tooth restoration
- e.max (Active Comparator): Restorations in e.max bonded to tooth substance by dual cure resin cement
  Interventions: Other: Ceramic tooth restoration

INTERVENTIONS:
Other: Ceramic tooth restoration — Dental restorations

SUMMARY:
This randomized clinical study aims to compare success and survival of two different ceramic tooth restoration materials. The hypothesis for the study is that fluoride treated zirconia will retain as good as lithium disilicate reinforced glass ceramic when cemented by the same resin cement.

One group of patients will receive a restoration in fluoride treated zirconia, the other group will receive a restoration in reinforced glass ceramic. All restorations will be cemented in the same manner. At 3, 6, 12 and 24 months the participants will be examined.

DETAILED DESCRIPTION:
A randomized controlled clinical study that aims to compare success and survival of potassium hydrogen difluoride (KHF2) etched zirconium dioxide and lithium disilicate reinforced glass ceramic cemented to molars/premolares using dual cure resin cement.

The null hypothesis for the study is that zirconium dioxide and lithium disilicate reinforced glass ceramic will retain equally good tooth substance when cemented with resin cement.

Participants are recruited from the student clinic at Faculty of Dentistry, University of Oslo. Patients who fulfill the inclusion criteria 1) age above 18, 2) require restoration on premolar/molar and 3) are able to come to treatment and recall, are informed about the study and invited to participate. Consent to participation are signed by the patient. At any time and for any reason participants can withdraw from the study.

Personal information will be registered in Service for Sensitive Data, which is a platform to collect, store, analyze and share sensitive data. An encoded research file will be kept separate from the patient journal.The content of this file will be patient journal number and classification of the restoration on a four level scale (Californian Dental Association - CDA) for each recall.

A randomizing tool will be used to decide which ceramic restoration each participant will receive. Treatment will be performed by one clinician. The tooth preparation will be with little retention, and preferably supragingival. For cementing the restorations a standardized protocol for a dual cure resin cement will be used.

Participants only have to pay for the dental technician expenses and will be the same amount regardless of type of ceramic.

Each participant will be examined at 3, 6, 12 and 24 months by a clinician different from the one who performed the treatment. The 4 level CDA classification will be used to characterise each restoration.

Each of the two treatment groups will consist of 20 participants. Significant results will be achieved with the approximate distribution across categories: Category 1: 19,9 %, category 2: 79,4 %, category 3: 4,6 %, category 4: 2,5 %

ELIGIBILITY:
Inclusion Criteria:

18 years or older In the need of treatment on molars or premolars Lives near by Oslo

-

Exclusion Criteria:

The patients that does not fulfill the inclusion criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  Restoration still retained to tooth
Loss of retention | 2 years
  Restoration not retained to tooth

SECONDARY OUTCOMES:
CDA-index: Romeo | 2 years
  Excellent: Surface smooth and glossy, no mismatch in color or shade
CDA-index: Sierra | 2 years
  Acceptable: SRO: Surface slightly rough or pitted, can be polished. SMM: slight mismatch in shade
CDA-index: Tango | 2 years
  Correct: TGI: surface glossy irregular, not subject to correction. TMM: mismatch between restoration and adjacent teeth outside normal range.
CDA-index: Victor | 2 years
  Replace: VSF: surface fractured. VGP: Gross porosities. VSD: shade in gross disharmony

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eirik Ellingsen, Professor, Study Chair — Faculty of Dentistry, Institute of Clinical Dentistry
Locations (1):
- Institute of Clinical Dentistry, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
After termination of the study other researchers may use the database for further research

REFERENCES:
- [Background] Ruyter EI, Vajeeston N, Knarvang T, Kvam K. A novel etching technique for surface treatment of zirconia ceramics to improve adhesion of resin-based luting cements. Acta Biomater Odontol Scand. 2017 Apr 14;3(1):36-46. doi: 10.1080/23337931.2017.1309658. eCollection 2017 Jan. PMID 28642930